CLINICAL TRIAL: NCT05049135
Title: Long Distance Diagnostics of Sleep Apnea With Objective Sleep Data From a Sensor-less Monitor - a Feasibility Study
Brief Title: Feasibility of a Sensor-less Sleep Monitor (Somnofy®) in Diagnosis and Follow-up in Obstructive Sleep Apnea.
Status: Completed | Type: Observational
Sponsor: Helse Nord-Trøndelag HF (Other)
Collaborators: Norwegian University of Science and Technology (Other); VitalThings (Industry)
Responsible Party: Sponsor
Other Study IDs: 200405; CIV-NO-21-08-037486 (Other: Eudamed)
Record Dates: First submitted 2021-09-09; First posted 2021-09-17 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Obstructive Sleep Apnea
Keywords: sleep monitor
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sleep apnea group: Patients with undiagnosed suspected sleep apnea who are referred to Levanger Hospital for respiratory polygraphy
  Interventions: Device: Somnofy® sleep monitor
- Control group: partners of patients with undiagnosed suspected sleep apnea who are referred to Levanger Hospital for respiratory polygraphy
  Interventions: Device: Somnofy® sleep monitor

INTERVENTIONS:
Device: Somnofy® sleep monitor — Registration of sleep score and apneas with radar sensor technology at time of primary investigation and 12 weeks after treatment initiation with continuous positive airway pressure (CPAP)
  Other Names: Respiratory polygraphy (NOXT3, ResMed AS)

SUMMARY:
To evaluate the feasibility of a sensor-less sleep monitor (Somnofy®) in diagnosis and follow-up in obstructive sleep apnea. The study will explore the monitor's usefulness in detection of apnea during sleep, and compare the data to standard diagnostic registrations.

DETAILED DESCRIPTION:
A single-center prospective feasibility study. The study device is Somnofy®, a sensor-less commercially available sleep monitor. The ability of the monitor to detect apneas or hypopneas based on ultra wideband radar technology will be evaluated. The Somnofy® radar data will be compared with the diagnostic data from the predicate polygraph device NOX-T3 and the OSAS event data from the Metronics AirView software from CPAP. Thus, it will be possible to assess if Somnofy® is able to detect the events registered from the diagnostic equipment. For patients started on Continous Positive Airway Pressure (CPAP) treatment, a new registration with Somnofy® will be performed 12 weeks after treatment initiation. The effect of obstructive sleep apnea on patient and partner reported outcomes before and after CPAP initiation will also be assessed through questionnaires and journals.

ELIGIBILITY:
Inclusion Criteria:

* referred to the pulmonology department in the participating hospital (Sykehuset Levanger) with suspected sleep apnea
* able to sign an informed consent

Exclusion Criteria:

* Pregnancy
* Serious disease which could affect ability to complete the study
* Complicated sleep disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patents with undiagnosed suspected sleep apnea who are referred to Levanger Hospital for respiratory polygraphy, and their partners
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-03-07 (Actual)

PRIMARY OUTCOMES:
Apnea/hypopnea index | 72 hours
  Apnea/hypopnea index defined as the number of apneas or hypopneas per hours of sleep

SECONDARY OUTCOMES:
Sleep score | 12 weeks
  Objective (AI-based) score of sleep quality from raw data from sleep monitor

CONTACTS AND LOCATIONS:
Overall Officials: Øystein Risa, PhD, Study Director — NTNU, Fac of Med and Health Sci, Dept of Circulation and Medical Imaging; Carl Platou, MD, Study Director — North Trøndelag Hospital Trust
Locations (1):
- Department of Pulmonology, Levanger Hospital, North Trøndelag Hospital Trust, Levanger, Norway